CLINICAL TRIAL: NCT07149506
Title: Efficacy of Oral or Topical Catechins vs. Placebo as an Adjuvant for the Prevention and Management of Radiation Dermatitis in Oncology Patients: a Randomized Trial
Brief Title: Oral or Topical Catechins for Radiation Dermatitis
Acronym: OCTOPUS-RD
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: CARLOS FRANCISCO SAAVEDRA GARCIA (Other)
Collaborators: Universidad de Guanajuato (Other); Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Sponsor-Investigator, CARLOS FRANCISCO SAAVEDRA GARCIA, Principal Investigator, Universidad de Guanajuato
Organization: Universidad de Guanajuato (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEI-038-2025; CI/HRAEB/024/2025 (Other: IMSS Bienestar)
Record Dates: First submitted 2025-08-06; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Radiation Dermatitis Acute; Radiation Dermatitis; Fibrosis; Skin
Keywords: Catechins; Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis; Fibrosis | interventions — Catechin; epigallocatechin gallate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Oral epicatechin prevention group (Experimental): Oral epicatechin at a dose of 50 mg orally every 12 hours, starting from the start of radiotherapy, considering that one dose should be taken 2.5 hours before radiotherapy.
  Interventions: Other: Epicatechin
- Oral placebo prevention group (Placebo Comparator): Microcrystalline cellulose at a dose of 50 mg orally every 12 hours, starting from the start of radiotherapy, considering that one dose should be taken 2.5 hours before radiotherapy.
  Interventions: Other: Microcrystalline Cellulose NF (placebo)
- Topical epigallocatechin-3 gallate (EGCG) prevention group (Experimental): EGCG 660 μmol/L solution will be applied 0.5mL/cm2, 3 times a day in the treatment area from the start of radiotherapy and up to 2 weeks after the end of radiotherapy.
  Interventions: Other: Epigallocatechin Gallate (EGCG)
- Topical placebo prevention group (Placebo Comparator): Application of 0.5 mL/cm2 of 0.9% saline solution to the treatment area, three times per day. This regimen should be followed from the onset of radiotherapy until two weeks post-radiotherapy.
  Interventions: Other: Saline (0.9% NaCl)
- Oral epicatechin treatment group (Experimental): Oral epicatechin at a dose of 50 mg orally every 12 hours from the development of grade 1 radiodermatitis, considering that one should be taken 2.5 hours before radiotherapy.
  Interventions: Other: Epicatechin
- Oral placebo treatment group (Placebo Comparator): Microcrystalline cellulose at a dose of 50 mg orally every 12 hours, starting from the development of grade 1 radiodermatitis, considering that a dose should be taken 2.5 hours before radiotherapy.
  Interventions: Other: Microcrystalline Cellulose NF (placebo)
- Topical EGCG treatment group (Experimental): A solution of epigallocatechin-3 gallate (EGCG) 660 μmol/L, 0.5 mL/cm2, will be applied 3 times a day to the area to be treated from the development of grade 1 radiodermatitis and up to 2 weeks after the end of radiotherapy.
  Interventions: Other: Epigallocatechin Gallate (EGCG)
- Topical placebo treatment group (Placebo Comparator): Application of 0.5 mL/cm2 of 0.9% saline solution to the treatment area, three times per day. This regimen should be followed from the development of grade 1 radiodermatitis until two weeks post-radiotherapy.
  Interventions: Other: Saline (0.9% NaCl)

INTERVENTIONS:
Other: Epicatechin — A comparison will be made between oral catechin (epicatechin) from two approaches: a preventive approach and a therapeutic approach.
  Arms: Oral epicatechin prevention group; Oral epicatechin treatment group
Other: Epigallocatechin Gallate (EGCG) — A comparison will be made between topical catechin (EGCG) from two approaches: a preventive approach and a therapeutic approach.
  Other Names: Epigallocatechin-3 Gallate
  Arms: Topical EGCG treatment group; Topical epigallocatechin-3 gallate (EGCG) prevention group
Other: Microcrystalline Cellulose NF (placebo) — A comparison will be made between oral placebo (microcrystalline cellulose) from two approaches: a preventive approach and a therapeutic approach.
  Other Names: Placebo
  Arms: Oral placebo prevention group; Oral placebo treatment group
Other: Saline (0.9% NaCl) — A comparison will be made between topical placebo (0.9% saline solution) from two approaches: a preventive approach and a therapeutic approach.
  Other Names: Placebo
  Arms: Topical placebo prevention group; Topical placebo treatment group

SUMMARY:
Introduction Radiation-induced dermatitis (RID), which includes both acute and chronic forms, affects up to 95% of patients undergoing radiation therapy. Despite its high incidence, there are currently no validated prevention and management recommendations specifically for the mexican population. Catechins, particularly epigallocatechin gallate and epicatechin, are emerging as a promising and readily accessible therapeutic option for radiation damage in skin and other organs, including conditions like esophagitis, intestinal injury, and mucositis.

Objective This study aims to evaluate the utility of oral or topical catechins in preventing and managing acute and chronic radiation-induced dermatitis in cancer patients, comparing their effectiveness against standard treatment.

Material and Methods

This will be a randomized, double-blind, phase III clinical trial with a longitudinal and comparative design. Patients will be allocated into two primary study groups: prevention (n=81) and treatment (n=81). Each group will be further divided into four treatment arms:

Epigallocatechin gallate (experimental aerosol)

Epicatechin (experimental capsule)

Saline control arm (aerosol)

Microcrystalline cellulose excipient control arm (capsule)

All participants across all groups will receive standard care. Study endpoints will include the assessment of utility, toxicity, quality of life, and cosmesis, using various validated scales and scores.

Ethics This study adheres to the principles outlined in the Helsinki Declaration (2024), the Nuremberg Code, and Mexico's General Health Law on health research. Given the wide therapeutic margin of the interventions, the study is classified as minimal risk.

Statistical Analysis To evaluate the efficacy of the intervention (specifically, the change in the risk of dermatitis and fibrosis), we will calculate the hazard ratio using Cox regression and compare it with the Log-Rank test. Additionally, both fixed and random effects models will be performed and compared using the likelihood ratio test.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of cancer.
* Complete blood count, blood chemistry, and liver function tests within normal ranges.
* Availability of an anatomopathological report.
* Aged between 18 and 75 years.
* Karnofsky performance status (KPS) score > 60 or an Eastern Cooperative Oncology Group (ECOG) performance status score < 3.
* Candidate for radiotherapy with a prescribed dose of ≥40 Gy or its biological equivalent (EQD2).
* Must provide written informed consent to participate in the study.
* Must be able to swallow capsules.
* Must meet one of the following cohort-specific criteria:

  1. Prevention cohort: No clinical evidence of dermatitis at the initiation of radiotherapy.
  2. Treatment cohort: Development of grade 1 dermatitis during radiotherapy, with symptom onset within the last 3 days.

Exclusion Criteria:

* Pregnant or lactating.
* Immunocompromised or on chronic therapy with immunosuppressive or immunomodulatory medications.
* History of chemical burns or unhealed wounds in the intended radiotherapy treatment area.
* Current diagnosis of skin cancer or a known diagnosis of a DNA repair gene defect.
* Prior radiotherapy to the area currently being treated.
* Known allergy to any of the study compounds.
* Currently receiving treatment with bortezomib, sunitinib, ticagrelor, or other antithrombotic agents.

Withdrawal Criteria:

* Adherence to the study intervention is less than 80%.
* Withdrawal of consent.
* Suspension of their radiotherapy sessions secondary to an acute infectious disease or the need for hospitalization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of chronic radiation fibrosis | A baseline RTOG scale evaluation is performed before the placebo or catechins treatment begins. Following treatment, primary measurements for fibrosis are taken during follow-up visits at 3 and 6 months post-radiotherapy.
  Chronic radiation dermatitis/fibrosis This condition is defined as an adverse skin reaction that occurs more than 90 days after the start of radiotherapy. It involves permanent structural changes to the skin, such as fibrosis and vascular atrophy. Fibrosis can increase the risk of poor wound healing, skin contractures, and pain.
  Radiation therapy oncology group (RTOG) scale The RTOG scale is a standardized tool used to grade late-stage radiation effects. For the purposes of this study, the presence of fibrosis is graded on an ordinal scale with a minimum value of 0 and a maximum value of 2. On this scale, a higher score indicates a worse outcome (more severe fibrosis).
Change in the radiation-induced skin reaction assessment scale (RISRAS) score | A baseline RISRAS scale evaluation is performed before the placebo or catechins treatment begins. Subsequent measurements are then taken up to week 7 during radiotherapy, and at 1 week and 2 weeks post-radiotherapy.
  The Radiation-Induced Skin Reaction Assessment Scale (RISRAS) measures the severity of skin reactions to radiotherapy. It combines a clinician's assessment of visible signs with the patient's self-reported symptoms. A higher score, with a maximum of 37.5 points, indicates a more severe reaction.
  Clinicians apply the RISRAS scale to assess the the severity of acute radiation dermatitis.
  The change from baseline will be compared between the catechin and placebo groups to determine the impact on symptom severity.

SECONDARY OUTCOMES:
Incidence of Adverse Events | A baseline CTCAE v5.0 scale evaluation is performed before the placebo or catechins treatment begins. Subsequent evaluations are then conducted up to week 7 during radiotherapy and again at 3 months post-radiotherapy.
  Outcome Measure Description:
  The frequency of adverse events, such as hepatic or hematological toxicity, will be quantified and compared between the catechin and placebo groups.
  Common Terminology Criteria for Adverse Events (CTCAE) v5.0 will be used as the standardized system for grading the severity of acute adverse events. For this study, the events will be graded on its 5-point scale, ranging from a minimum of Grade 1 (mild) to a maximum of Grade 5 (death related to the adverse event). A higher score on this scale indicates a worse outcome.
Dermatological Quality of Life | The measurement will be taken at baseline (before the placebo or catechins treatment begins), weekly up to week 7 during radiotherapy, and at 3 and 6 months post-radiotherapy.
  Outcome Measure Description:
  The skin-related quality of life (QoL) will be determined and compared among patients in the different treatment groups. It will be evaluated using the Skindex-16 questionnaire, a validated 16-item tool that measures skin-specific QoL across three domains: symptoms, emotions, and functioning. The questionnaire has a minimum score of 0 and a maximum score of 100. On this scale, a higher score indicates a worse QoL.
Cumulative radiation dose at onset of grade ≥2 dermatitis | Measurements are taken throughout radiotherapy, up to week 7, with additional assessments at 1 and 2 weeks after the radiotherapy period.
  The total radiation dose (in Gray - Gy) delivered to the skin at the precise moment the first clinical signs of grade 2 (or higher) radiation dermatitis are observed, as assessed by the radiation-induced skin reaction assessment scale (RISRAS).
  Interpretation: A higher cumulative dose (Gy) indicates a better outcome. It signifies greater radioprotection from the intervention, allowing the patient to tolerate more radiotherapy before experiencing significant skin toxicity.
  Unit of measure: Gray (Gy).
Cosmetic Outcome | Photographs will be taken at three key points: Baseline, before the placebo or catechins treatment begins. During radiotherapy, specifically at weeks 1 and 3 of treatment. Post-radiotherapy, at both 3 and 6 months after treatment.
  The cosmetic results of the skin in the treated area will be evaluated. This will be measured objectively using serial photographs. The photographs will be analyzed quantitatively with ImageJ software (National Institutes of Health, Bethesda, MD) to measure and compare changes in skin appearance (e.g., erythema, pigmentation, texture) between the catechin and placebo groups.
  Interpretation of results:
  Objective quantitative analysis: A statistically significant improvement in the quantitative skin appearance metrics (e.g., reduced erythema, improved homogeneity) in the catechin group compared to the placebo group at the post-radiotherapy time points indicates a better cosmetic outcome.
  A lack of significant difference or worse metrics in the catechin group would indicate no benefit or a worse outcome, respectively.
Duration of grade ≥2 dermatitis | Measurements are taken throughout radiotherapy, up to week 7, with additional assessments at 1 and 2 weeks after the radiotherapy period.
  The length of time (in days) that the radiation dermatitis persists at a severity of Grade 2 or higher, from its onset until its resolution to grade 1 or lower, as measured by the radiation-induced skin reaction assessment scale (RISRAS).
  Interpretation: A shorter duration (fewer days) indicates a better outcome. It signifies a faster recovery and resolution of the skin adverse event, potentially improving patient quality of life and reducing treatment interruptions.
  Unit of measure: Days.
Percentage of Affected Skin Area by Radiation Dermatitis | Baseline, week 1, and week 3 of radiotherapy.
  Standardized photographs of the irradiated area will be taken and analyzed using ImageJ® software to objectively quantify the percentage of skin affected by dermatitis. This objective measurement will be compared between the catechin and placebo groups.
  Unit of measure: Percentage (%).
  A higher percentage of affected skin indicates a more severe cutaneous reaction to radiation, while a lower percentage suggests a better clinical outcome and greater radioprotection.

OTHER OUTCOMES:
Compare the efficacy of a topical epigallocatechin-3-gallate (EGCG) aerosol versus an oral epicatechin (Epi) capsule | The efficacy comparison of topical epigallocatechin gallate versus oral epicatechin will be conducted at the following times: at baseline (before administration), at week 7, 1 week post-radiotherapy, and 2 weeks post-radiotherapy.
  The efficacy of topical versus oral administration routes will be compared using mixed-effects models to account for repeated measures and variability within subjects.
  Statistical Method: A Wald test will be applied to the coefficient of the administration route term in the mixed model to determine if there is a statistically significant difference in efficacy between the two treatment groups.
  Interpretation of results: A statistically significant Wald test result (p < 0.05) for the administration route coefficient indicates a significant difference in efficacy between topical and oral treatments. The direction and magnitude of the coefficient will determine which route is superior. A non-significant result suggests no detectable difference in efficacy between the two administration routes.
Explore the 6-month event-free survival (EFS) of the study groups | 6 months after radiotherapy concludes.
  Patient status is monitored throughout the study's follow-up period to determine the date of any event, defined as disease progression, cancer recurrence, or death from any cause.
  Statistical Method: EFS will be analyzed using Kaplan-Meier curves to visually compare the probability of remaining event-free between the study groups over the 6-month follow-up period. The log-rank test will be used to assess statistical significance.
  Interpretation of Results: A higher probability of event-free survival (i.e., a Kaplan-Meier curve that remains higher for longer) in the catechin group compared to the placebo group indicates a better clinical outcome. A statistically significant improvement (p < 0.05) would suggest that the intervention reduces the risk of disease progression, recurrence, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Palacios, MD; PhD; MMSc; genetics, Study Director
Locations (1):
- HRAEB, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available immediately following publication of the manuscript reporting the primary results (Start Date: March 2027) and will remain accessible until March 2032 (End Date: March 2032).
Access Criteria: De-identified IPD and supporting documents will be accessible to qualified researchers who provide a methodologically sound research proposal approved by an independent Data Access Committee (DAC). Requestors must also provide IRB/IEC approval for their proposed analysis and sign a Data Use Agreement (DUA) committing to data privacy, confidentiality, and use solely for the approved purpose.
  Requests should be submitted via email to comite.investigación@hraeb.gob.mx. Approved data will be transferred securely using encrypted methods

REFERENCES:
- [Background] Rey JL, Felix H, De Bary JB, Haller L. Ceftriaxone for treatment of severe infections in peripheral health centers in Africa. Chemioterapia. 1987 Jun;6(2 Suppl):382-3. No abstract available. PMID 2855614
- [Background] Masek P, Winklerova S. [Fluorescein and its adverse effects]. Cesk Oftalmol. 1989 Sep;45(5):362-4. Czech. PMID 2805111
- [Background] Fraser IE. Proteins of keratin and their synthesis. II. Incorporation of [35S]cystine into prekeratin and keratin proteins. Aust J Biol Sci. 1969 Feb;22(1):231-8. No abstract available. PMID 5783763
- [Background] Vollmann J, Winau R. Informed consent in human experimentation before the Nuremberg code. BMJ. 1996 Dec 7;313(7070):1445-9. doi: 10.1136/bmj.313.7070.1445. PMID 8973233
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: Ethical Principles for Medical Research Involving Human Participants. JAMA. 2025 Jan 7;333(1):71-74. doi: 10.1001/jama.2024.21972. PMID 39425955
- [Background] Hopewell S, Chan AW, Collins GS, Hrobjartsson A, Moher D, Schulz KF, Tunn R, Aggarwal R, Berkwits M, Berlin JA, Bhandari N, Butcher NJ, Campbell MK, Chidebe RCW, Elbourne D, Farmer A, Fergusson DA, Golub RM, Goodman SN, Hoffmann TC, Ioannidis JPA, Kahan BC, Knowles RL, Lamb SE, Lewis S, Loder E, Offringa M, Ravaud P, Richards DP, Rockhold FW, Schriger DL, Siegried NL, Staniszewska S, Taylor RS, Thabane L, Torgerson D, Vohra S, White IR, Boutron I. CONSORT 2025 statement: Updated guideline for reporting randomised trials. PLoS Med. 2025 Apr 14;22(4):e1004587. doi: 10.1371/journal.pmed.1004587. eCollection 2025 Apr. PMID 40228477
- [Background] Wooding H, Yan J, Yuan L, Chyou TY, Gao S, Ward I, Herst PM. The effect of Mepitel Film on acute radiation-induced skin reactions in head and neck cancer patients: a feasibility study. Br J Radiol. 2018 Jan;91(1081):20170298. doi: 10.1259/bjr.20170298. Epub 2017 Nov 8. PMID 29072852
- [Background] Robijns J, Censabella S, Claes S, Pannekoeke L, Busse L, Colson D, Kaminski I, Bulens P, Maes A, Noe L, Brosens M, Timmermans A, Lambrichts I, Somers V, Mebis J. Prevention of acute radiodermatitis by photobiomodulation: A randomized, placebo-controlled trial in breast cancer patients (TRANSDERMIS trial). Lasers Surg Med. 2018 Feb 10. doi: 10.1002/lsm.22804. Online ahead of print. PMID 29427390
- [Background] Yu Z, Samavat H, Dostal AM, Wang R, Torkelson CJ, Yang CS, Butler LM, Kensler TW, Wu AH, Kurzer MS, Yuan JM. Effect of Green Tea Supplements on Liver Enzyme Elevation: Results from a Randomized Intervention Study in the United States. Cancer Prev Res (Phila). 2017 Oct;10(10):571-579. doi: 10.1158/1940-6207.CAPR-17-0160. Epub 2017 Aug 1. PMID 28765194
- [Background] EFSA Panel on Food Additives and Nutrient Sources added to Food (ANS); Younes M, Aggett P, Aguilar F, Crebelli R, Dusemund B, Filipic M, Frutos MJ, Galtier P, Gott D, Gundert-Remy U, Lambre C, Leblanc JC, Lillegaard IT, Moldeus P, Mortensen A, Oskarsson A, Stankovic I, Waalkens-Berendsen I, Woutersen RA, Andrade RJ, Fortes C, Mosesso P, Restani P, Arcella D, Pizzo F, Smeraldi C, Wright M. Scientific opinion on the safety of green tea catechins. EFSA J. 2018 Apr 18;16(4):e05239. doi: 10.2903/j.efsa.2018.5239. eCollection 2018 Apr. PMID 32625874
- [Background] Zhao H, Zhu W, Jia L, Sun X, Chen G, Zhao X, Li X, Meng X, Kong L, Xing L, Yu J. Phase I study of topical epigallocatechin-3-gallate (EGCG) in patients with breast cancer receiving adjuvant radiotherapy. Br J Radiol. 2016;89(1058):20150665. doi: 10.1259/bjr.20150665. Epub 2015 Nov 26. PMID 26607642
- [Background] Zhu W, Jia L, Chen G, Zhao H, Sun X, Meng X, Zhao X, Xing L, Yu J, Zheng M. Epigallocatechin-3-gallate ameliorates radiation-induced acute skin damage in breast cancer patients undergoing adjuvant radiotherapy. Oncotarget. 2016 Jul 26;7(30):48607-48613. doi: 10.18632/oncotarget.9495. PMID 27224910
- [Background] Landis-Piwowar K, Chen D, Foldes R, Chan TH, Dou QP. Novel epigallocatechin gallate analogs as potential anticancer agents: a patent review (2009 - present). Expert Opin Ther Pat. 2013 Feb;23(2):189-202. doi: 10.1517/13543776.2013.743993. Epub 2012 Dec 12. PMID 23230990
- [Background] Xu FW, Lv YL, Zhong YF, Xue YN, Wang Y, Zhang LY, Hu X, Tan WQ. Beneficial Effects of Green Tea EGCG on Skin Wound Healing: A Comprehensive Review. Molecules. 2021 Oct 11;26(20):6123. doi: 10.3390/molecules26206123. PMID 34684703
- [Background] Hwang Y, Chang B, Kim T, Kim S. Ameliorative effects of green tea extract from tannase digests on house dust mite antigen-induced atopic dermatitis-like lesions in NC/Nga mice. Arch Dermatol Res. 2019 Mar;311(2):109-120. doi: 10.1007/s00403-018-01886-6. Epub 2019 Jan 7. PMID 30617657
- [Background] Chamcheu JC, Siddiqui IA, Adhami VM, Esnault S, Bharali DJ, Babatunde AS, Adame S, Massey RJ, Wood GS, Longley BJ, Mousa SA, Mukhtar H. Chitosan-based nanoformulated (-)-epigallocatechin-3-gallate (EGCG) modulates human keratinocyte-induced responses and alleviates imiquimod-induced murine psoriasiform dermatitis. Int J Nanomedicine. 2018 Jul 20;13:4189-4206. doi: 10.2147/IJN.S165966. eCollection 2018. PMID 30057446
- [Background] Wang ZT, Xue Y, Sun H, Zhang Z, Tang ZJ, Liu SB, Cai WM. Effect of tea polyphenols on the oral and intravenous pharmacokinetics of ticagrelor in rats and its in vitro metabolism. J Food Sci. 2020 Apr;85(4):1285-1291. doi: 10.1111/1750-3841.15096. Epub 2020 Mar 10. PMID 32157685
- [Background] Ge J, Tan BX, Chen Y, Yang L, Peng XC, Li HZ, Lin HJ, Zhao Y, Wei M, Cheng K, Li LH, Dong H, Gao F, He JP, Wu Y, Qiu M, Zhao YL, Su JM, Hou JM, Liu JY. Interaction of green tea polyphenol epigallocatechin-3-gallate with sunitinib: potential risk of diminished sunitinib bioavailability. J Mol Med (Berl). 2011 Jun;89(6):595-602. doi: 10.1007/s00109-011-0737-3. Epub 2011 Feb 18. PMID 21331509
- [Background] Golden EB, Lam PY, Kardosh A, Gaffney KJ, Cadenas E, Louie SG, Petasis NA, Chen TC, Schonthal AH. Green tea polyphenols block the anticancer effects of bortezomib and other boronic acid-based proteasome inhibitors. Blood. 2009 Jun 4;113(23):5927-37. doi: 10.1182/blood-2008-07-171389. Epub 2009 Feb 3. PMID 19190249
- [Background] Yen C, Zhao F, Yu Z, Zhu X, Li CG. Interactions Between Natural Products and Tamoxifen in Breast Cancer: A Comprehensive Literature Review. Front Pharmacol. 2022 Jun 2;13:847113. doi: 10.3389/fphar.2022.847113. eCollection 2022. PMID 35721162
- [Background] Esmaeili MA. Combination of siRNA-directed gene silencing with epigallocatechin-3-gallate (EGCG) reverses drug resistance in human breast cancer cells. J Chem Biol. 2015 Aug 8;9(1):41-52. doi: 10.1007/s12154-015-0144-2. eCollection 2016 Jan. PMID 26855680
- [Background] La X, Zhang L, Li Z, Li H, Yang Y. (-)-Epigallocatechin Gallate (EGCG) Enhances the Sensitivity of Colorectal Cancer Cells to 5-FU by Inhibiting GRP78/NF-kappaB/miR-155-5p/MDR1 Pathway. J Agric Food Chem. 2019 Mar 6;67(9):2510-2518. doi: 10.1021/acs.jafc.8b06665. Epub 2019 Feb 20. PMID 30741544
- [Background] Chang CM, Chang PY, Tu MG, Lu CC, Kuo SC, Amagaya S, Lee CY, Jao HY, Chen MY, Yang JS. Epigallocatechin gallate sensitizes CAL-27 human oral squamous cell carcinoma cells to the anti-metastatic effects of gefitinib (Iressa) via synergistic suppression of epidermal growth factor receptor and matrix metalloproteinase-2. Oncol Rep. 2012 Nov;28(5):1799-807. doi: 10.3892/or.2012.1991. Epub 2012 Aug 24. PMID 22923287
- [Background] Zhou H, Fu LX, Li L, Chen YY, Zhu HQ, Zhou JL, Lv MX, Gan RZ, Zhang XX, Liang G. The epigallocatechin gallate derivative Y6 reduces the cardiotoxicity and enhances the efficacy of daunorubicin against human hepatocellular carcinoma by inhibiting carbonyl reductase 1 expression. J Ethnopharmacol. 2020 Oct 28;261:113118. doi: 10.1016/j.jep.2020.113118. Epub 2020 Jul 1. PMID 32621953
- [Background] Lang M, Henson R, Braconi C, Patel T. Epigallocatechin-gallate modulates chemotherapy-induced apoptosis in human cholangiocarcinoma cells. Liver Int. 2009 May;29(5):670-7. doi: 10.1111/j.1478-3231.2009.01984.x. Epub 2009 Feb 17. PMID 19226332
- [Background] Shervington A, Pawar V, Menon S, Thakkar D, Patel R. The sensitization of glioma cells to cisplatin and tamoxifen by the use of catechin. Mol Biol Rep. 2009 May;36(5):1181-6. doi: 10.1007/s11033-008-9295-3. Epub 2008 Jun 26. PMID 18581255
- [Background] Lee TC, Cheng IC, Shue JJ, Wang TC. Cytotoxicity of arsenic trioxide is enhanced by (-)-epigallocatechin-3-gallate via suppression of ferritin in cancer cells. Toxicol Appl Pharmacol. 2011 Jan 1;250(1):69-77. doi: 10.1016/j.taap.2010.10.005. Epub 2010 Oct 13. PMID 20950636
- [Background] Sanchez Y, Calle C, de Blas E, Aller P. Modulation of arsenic trioxide-induced apoptosis by genistein and functionally related agents in U937 human leukaemia cells. Regulation by ROS and mitogen-activated protein kinases. Chem Biol Interact. 2009 Nov 10;182(1):37-44. doi: 10.1016/j.cbi.2009.08.015. Epub 2009 Aug 29. PMID 19720055
- [Background] Wang L, Li P, Feng K. EGCG adjuvant chemotherapy: Current status and future perspectives. Eur J Med Chem. 2023 Mar 15;250:115197. doi: 10.1016/j.ejmech.2023.115197. Epub 2023 Feb 10. PMID 36780831
- [Background] Zhao H, Zhu W, Xie P, Li H, Zhang X, Sun X, Yu J, Xing L. A phase I study of concurrent chemotherapy and thoracic radiotherapy with oral epigallocatechin-3-gallate protection in patients with locally advanced stage III non-small-cell lung cancer. Radiother Oncol. 2014 Jan;110(1):132-6. doi: 10.1016/j.radonc.2013.10.014. Epub 2014 Jan 17. PMID 24444526
- [Background] Shin DM, Nannapaneni S, Patel MR, Shi Q, Liu Y, Chen Z, Chen AY, El-Deiry MW, Beitler JJ, Steuer CE, Roser SM, Klein AM, Owonikoko TK, Ramalingam SS, Khuri FR, Chen ZG, Saba NF. Phase Ib Study of Chemoprevention with Green Tea Polyphenon E and Erlotinib in Patients with Advanced Premalignant Lesions (APL) of the Head and Neck. Clin Cancer Res. 2020 Nov 15;26(22):5860-5868. doi: 10.1158/1078-0432.CCR-20-2276. Epub 2020 Sep 17. PMID 32943457
- [Background] Zhu W, Mei H, Jia L, Zhao H, Li X, Meng X, Zhao X, Xing L, Yu J. Epigallocatechin-3-gallate mouthwash protects mucosa from radiation-induced mucositis in head and neck cancer patients: a prospective, non-randomised, phase 1 trial. Invest New Drugs. 2020 Aug;38(4):1129-1136. doi: 10.1007/s10637-019-00871-8. Epub 2019 Nov 7. PMID 31701429
- [Background] Zhang G, Wang Y, Zhang Y, Wan X, Li J, Liu K, Wang F, Liu K, Liu Q, Yang C, Yu P, Huang Y, Wang S, Jiang P, Qu Z, Luan J, Duan H, Zhang L, Hou A, Jin S, Hsieh TC, Wu E. Anti-cancer activities of tea epigallocatechin-3-gallate in breast cancer patients under radiotherapy. Curr Mol Med. 2012 Feb;12(2):163-76. doi: 10.2174/156652412798889063. PMID 22280355
- [Background] Li X, Xing L, Zhang Y, Xie P, Zhu W, Meng X, Wang Y, Kong L, Zhao H, Yu J. Phase II Trial of Epigallocatechin-3-Gallate in Acute Radiation-Induced Esophagitis for Esophagus Cancer. J Med Food. 2020 Jan;23(1):43-49. doi: 10.1089/jmf.2019.4445. Epub 2019 Nov 20. PMID 31747326
- [Background] Zhao H, Xie P, Li X, Zhu W, Sun X, Sun X, Chen X, Xing L, Yu J. A prospective phase II trial of EGCG in treatment of acute radiation-induced esophagitis for stage III lung cancer. Radiother Oncol. 2015 Mar;114(3):351-6. doi: 10.1016/j.radonc.2015.02.014. Epub 2015 Mar 10. PMID 25769379
- [Background] Lu H, Xie L, Guo L, Gu X, Zhu R, Yang Y, Tang F, Li M, Liu C, Wang D, Li M, Tian Y, Cai S. EGCG protects intestines of mice and pelvic cancer patients against radiation injury via the gut microbiota/D-tagatose/AMPK axis. Radiother Oncol. 2025 Jan;202:110608. doi: 10.1016/j.radonc.2024.110608. Epub 2024 Oct 31. PMID 39486483
- [Background] Kang Y, Xiong Y, Lu B, Wang Y, Zhang D, Feng J, Chen L, Zhang Z. Application of In Situ Mucoadhesive Hydrogel with Anti-Inflammatory and Pro-Repairing Dual Properties for the Treatment of Chemotherapy-Induced Oral Mucositis. ACS Appl Mater Interfaces. 2024 Jul 17;16(28):35949-35963. doi: 10.1021/acsami.4c03217. Epub 2024 Jul 6. PMID 38970482
- [Background] Kapoor MP, Sugita M, Fukuzawa Y, Timm D, Ozeki M, Okubo T. Green Tea Catechin Association with Ultraviolet Radiation-Induced Erythema: A Systematic Review and Meta-Analysis. Molecules. 2021 Jun 17;26(12):3702. doi: 10.3390/molecules26123702. PMID 34204433
- [Background] Najera N, Ortiz-Flores M, Perez-Duran J, Reyes-Munoz E, Romo-Yanez J, Ortiz-Luna G, Villarreal F, Meaney E, Ceballos G, Montoya-Estrada A. Improving Cardiovascular Risk in Postmenopausal Women with an (-)-Epicatechin-Based Nutraceutical: A Randomly Assigned, Double-Blind vs. Placebo, Proof-of-Concept Trial. J Clin Med. 2023 Dec 29;13(1):195. doi: 10.3390/jcm13010195. PMID 38202201
- [Background] Gutierrez-Salmean G, Meaney E, Lanaspa MA, Cicerchi C, Johnson RJ, Dugar S, Taub P, Ramirez-Sanchez I, Villarreal F, Schreiner G, Ceballos G. A randomized, placebo-controlled, double-blind study on the effects of (-)-epicatechin on the triglyceride/HDLc ratio and cardiometabolic profile of subjects with hypertriglyceridemia: Unique in vitro effects. Int J Cardiol. 2016 Nov 15;223:500-506. doi: 10.1016/j.ijcard.2016.08.158. Epub 2016 Aug 8. PMID 27552564
- [Background] Zhao H, Zhu W, Zhao X, Li X, Zhou Z, Zheng M, Meng X, Kong L, Zhang S, He D, Xing L, Yu J. Efficacy of Epigallocatechin-3-Gallate in Preventing Dermatitis in Patients With Breast Cancer Receiving Postoperative Radiotherapy: A Double-Blind, Placebo-Controlled, Phase 2 Randomized Clinical Trial. JAMA Dermatol. 2022 Jul 1;158(7):779-786. doi: 10.1001/jamadermatol.2022.1736. PMID 35648426
- [Background] Xie J, Jia L, Xie P, Yin X, Zhu W, Zhao H, Wang X, Meng X, Xing L, Zhao H, Li X. Efficacy and safety of epigallocatechin-3-gallate in treatment acute severe dermatitis in patients with cancer receiving radiotherapy: a phase I clinical trial. Sci Rep. 2023 Aug 24;13(1):13865. doi: 10.1038/s41598-023-40881-4. PMID 37620508
- [Background] Arts IC, Hollman PC, Kromhout D. Chocolate as a source of tea flavonoids. Lancet. 1999 Aug 7;354(9177):488. doi: 10.1016/S0140-6736(99)02267-9. PMID 10465183
- [Background] Xicota L, Rodriguez-Morato J, Dierssen M, de la Torre R. Potential Role of (-)-Epigallocatechin-3-Gallate (EGCG) in the Secondary Prevention of Alzheimer Disease. Curr Drug Targets. 2017;18(2):174-195. doi: 10.2174/1389450116666150825113655. PMID 26302801
- [Background] Fernando WMADB, Somaratne G, Goozee KG, Williams S, Singh H, Martins RN. Diabetes and Alzheimer's Disease: Can Tea Phytochemicals Play a Role in Prevention? J Alzheimers Dis. 2017;59(2):481-501. doi: 10.3233/JAD-161200. PMID 28582855
- [Background] Mandel S, Maor G, Youdim MB. Iron and alpha-synuclein in the substantia nigra of MPTP-treated mice: effect of neuroprotective drugs R-apomorphine and green tea polyphenol (-)-epigallocatechin-3-gallate. J Mol Neurosci. 2004;24(3):401-16. doi: 10.1385/JMN:24:3:401. PMID 15655262
- [Background] Jiang S, Huang C, Zheng G, Yi W, Wu B, Tang J, Liu X, Huang B, Wu D, Yan T, Li M, Wan C, Cai Y. EGCG Inhibits Proliferation and Induces Apoptosis Through Downregulation of SIRT1 in Nasopharyngeal Carcinoma Cells. Front Nutr. 2022 Apr 25;9:851972. doi: 10.3389/fnut.2022.851972. eCollection 2022. PMID 35548580
- [Background] Cai S, Xie LW, Xu JY, Zhou H, Yang C, Tang LF, Tian Y, Li M. (-)-Epigallocatechin-3-Gallate (EGCG) Modulates the Composition of the Gut Microbiota to Protect Against Radiation-Induced Intestinal Injury in Mice. Front Oncol. 2022 Apr 11;12:848107. doi: 10.3389/fonc.2022.848107. eCollection 2022. PMID 35480105
- [Background] Kim SR, Seong KJ, Kim WJ, Jung JY. Epigallocatechin Gallate Protects against Hypoxia-Induced Inflammation in Microglia via NF-kappaB Suppression and Nrf-2/HO-1 Activation. Int J Mol Sci. 2022 Apr 4;23(7):4004. doi: 10.3390/ijms23074004. PMID 35409364
- [Background] Spencer JP, Schroeter H, Kuhnle G, Srai SK, Tyrrell RM, Hahn U, Rice-Evans C. Epicatechin and its in vivo metabolite, 3'-O-methyl epicatechin, protect human fibroblasts from oxidative-stress-induced cell death involving caspase-3 activation. Biochem J. 2001 Mar 15;354(Pt 3):493-500. doi: 10.1042/0264-6021:3540493. PMID 11237853
- [Background] Suzuki J, Ogawa M, Futamatsu H, Kosuge H, Sagesaka YM, Isobe M. Tea catechins improve left ventricular dysfunction, suppress myocardial inflammation and fibrosis, and alter cytokine expression in rat autoimmune myocarditis. Eur J Heart Fail. 2007 Feb;9(2):152-9. doi: 10.1016/j.ejheart.2006.05.007. Epub 2006 Jul 10. PMID 16829193
- [Background] Bhardwaj P, Khanna D. Green tea catechins: defensive role in cardiovascular disorders. Chin J Nat Med. 2013 Jul;11(4):345-53. doi: 10.1016/S1875-5364(13)60051-5. PMID 23845542
- [Background] Schiffrin EL. A critical review of the role of endothelial factors in the pathogenesis of hypertension. J Cardiovasc Pharmacol. 2001 Nov;38 Suppl 2:S3-6. doi: 10.1097/00005344-200111002-00002. PMID 11811373
- [Background] Galley HF, Webster NR. Physiology of the endothelium. Br J Anaesth. 2004 Jul;93(1):105-13. doi: 10.1093/bja/aeh163. Epub 2004 Apr 30. PMID 15121728
- [Background] Hu B, Pan C, Sun Y, Hou Z, Ye H, Zeng X. Optimization of fabrication parameters to produce chitosan-tripolyphosphate nanoparticles for delivery of tea catechins. J Agric Food Chem. 2008 Aug 27;56(16):7451-8. doi: 10.1021/jf801111c. Epub 2008 Jul 16. PMID 18627163
- [Background] Rashidinejad A, Birch EJ, Everett DW. A novel functional full-fat hard cheese containing liposomal nanoencapsulated green tea catechins: manufacture and recovery following simulated digestion. Food Funct. 2016 Jul 13;7(7):3283-94. doi: 10.1039/c6fo00354k. PMID 27374326
- [Background] Rashidinejad A, Birch EJ, Sun-Waterhouse D, Everett DW. Delivery of green tea catechin and epigallocatechin gallate in liposomes incorporated into low-fat hard cheese. Food Chem. 2014 Aug 1;156:176-83. doi: 10.1016/j.foodchem.2014.01.115. Epub 2014 Feb 6. PMID 24629955
- [Background] Rashidinejad A, Boostani S, Babazadeh A, Rehman A, Rezaei A, Akbari-Alavijeh S, Shaddel R, Jafari SM. Opportunities and challenges for the nanodelivery of green tea catechins in functional foods. Food Res Int. 2021 Apr;142:110186. doi: 10.1016/j.foodres.2021.110186. Epub 2021 Feb 1. PMID 33773663
- [Background] Wang R, Zhou W, Wen RA. Kinetic study of the thermal stability of tea catechins in aqueous systems using a microwave reactor. J Agric Food Chem. 2006 Aug 9;54(16):5924-32. doi: 10.1021/jf0611419. PMID 16881696
- [Background] Zeng J, Xu H, Cai Y, Xuan Y, Liu J, Gao Y, Luan Q. The Effect of Ultrasound, Oxygen and Sunlight on the Stability of (-)-Epigallocatechin Gallate. Molecules. 2018 Sep 18;23(9):2394. doi: 10.3390/molecules23092394. PMID 30231585
- [Background] Feng WY. Metabolism of green tea catechins: an overview. Curr Drug Metab. 2006 Oct;7(7):755-809. doi: 10.2174/138920006778520552. PMID 17073579
- [Background] Barnett CF, Moreno-Ulloa A, Shiva S, Ramirez-Sanchez I, Taub PR, Su Y, Ceballos G, Dugar S, Schreiner G, Villarreal F. Pharmacokinetic, partial pharmacodynamic and initial safety analysis of (-)-epicatechin in healthy volunteers. Food Funct. 2015 Mar;6(3):824-33. doi: 10.1039/c4fo00596a. PMID 25598082
- [Background] Youn HS, Lee JY, Saitoh SI, Miyake K, Kang KW, Choi YJ, Hwang DH. Suppression of MyD88- and TRIF-dependent signaling pathways of Toll-like receptor by (-)-epigallocatechin-3-gallate, a polyphenol component of green tea. Biochem Pharmacol. 2006 Sep 28;72(7):850-9. doi: 10.1016/j.bcp.2006.06.021. Epub 2006 Aug 4. PMID 16890209
- [Background] Bors W, Heller W, Michel C, Saran M. Flavonoids as antioxidants: determination of radical-scavenging efficiencies. Methods Enzymol. 1990;186:343-55. doi: 10.1016/0076-6879(90)86128-i. No abstract available. PMID 2172711
- [Background] Fan FY, Sang LX, Jiang M. Catechins and Their Therapeutic Benefits to Inflammatory Bowel Disease. Molecules. 2017 Mar 19;22(3):484. doi: 10.3390/molecules22030484. PMID 28335502
- [Background] Fraga CG, Galleano M, Verstraeten SV, Oteiza PI. Basic biochemical mechanisms behind the health benefits of polyphenols. Mol Aspects Med. 2010 Dec;31(6):435-45. doi: 10.1016/j.mam.2010.09.006. Epub 2010 Sep 18. PMID 20854840
- [Background] Babu PV, Liu D. Green tea catechins and cardiovascular health: an update. Curr Med Chem. 2008;15(18):1840-50. doi: 10.2174/092986708785132979. PMID 18691042
- [Background] Cabrera C, Artacho R, Gimenez R. Beneficial effects of green tea--a review. J Am Coll Nutr. 2006 Apr;25(2):79-99. doi: 10.1080/07315724.2006.10719518. PMID 16582024
- [Background] Braicu C, Ladomery MR, Chedea VS, Irimie A, Berindan-Neagoe I. The relationship between the structure and biological actions of green tea catechins. Food Chem. 2013 Dec 1;141(3):3282-9. doi: 10.1016/j.foodchem.2013.05.122. Epub 2013 Jun 4. PMID 23871088
- [Background] Bernatoniene J, Kopustinskiene DM. The Role of Catechins in Cellular Responses to Oxidative Stress. Molecules. 2018 Apr 20;23(4):965. doi: 10.3390/molecules23040965. PMID 29677167
- [Background] Elbaz HA, Lee I, Antwih DA, Liu J, Huttemann M, Zielske SP. Epicatechin stimulates mitochondrial activity and selectively sensitizes cancer cells to radiation. PLoS One. 2014 Feb 6;9(2):e88322. doi: 10.1371/journal.pone.0088322. eCollection 2014. PMID 24516636
- [Background] Parshad R, Sanford KK, Price FM, Steele VE, Tarone RE, Kelloff GJ, Boone CW. Protective action of plant polyphenols on radiation-induced chromatid breaks in cultured human cells. Anticancer Res. 1998 Sep-Oct;18(5A):3263-6. PMID 9858893
- [Background] Branda RF, Blickensderfer DB. Folate deficiency increases genetic damage caused by alkylating agents and gamma-irradiation in Chinese hamster ovary cells. Cancer Res. 1993 Nov 15;53(22):5401-8. PMID 8221678
- [Background] Umegaki K, Uramoto H, Suzuki J, Esashi T. Feeding mice palm carotene prevents DNA damage in bone marrow and reduction of peripheral leukocyte counts, and enhances survival following X-ray irradiation. Carcinogenesis. 1997 Oct;18(10):1943-7. doi: 10.1093/carcin/18.10.1943. PMID 9364004
- [Background] Harapanhalli RS, Yaghmai V, Giuliani D, Howell RW, Rao DV. Antioxidant effects of vitamin C in mice following X-irradiation. Res Commun Mol Pathol Pharmacol. 1996 Dec;94(3):271-87. PMID 9029674
- [Background] Yoshimura M, Kashiba M, Oka J, Sugisawa A, Umegaki K. Vitamin E prevents increase in oxidative damage to lipids and DNA in liver of ODS rats given total body X-ray irradiation. Free Radic Res. 2002 Jan;36(1):107-12. doi: 10.1080/10715760210166. PMID 11999697
- [Background] MacBride SK, Wells ME, Hornsby C, Sharp L, Finnila K, Downie L. A case study to evaluate a new soft silicone dressing, Mepilex Lite, for patients with radiation skin reactions. Cancer Nurs. 2008 Jan-Feb;31(1):E8-14. doi: 10.1097/01.NCC.0000305680.06143.39. PMID 18176123
- [Background] Shin YS, Shin HA, Kang SU, Kim JH, Oh YT, Park KH, Kim CH. Effect of epicatechin against radiation-induced oral mucositis: in vitro and in vivo study. PLoS One. 2013 Jul 18;8(7):e69151. doi: 10.1371/journal.pone.0069151. Print 2013. PMID 23874895
- [Background] Hoeller U, Tribius S, Kuhlmey A, Grader K, Fehlauer F, Alberti W. Increasing the rate of late toxicity by changing the score? A comparison of RTOG/EORTC and LENT/SOMA scores. Int J Radiat Oncol Biol Phys. 2003 Mar 15;55(4):1013-8. doi: 10.1016/s0360-3016(02)04202-5. PMID 12605981
- [Background] Gupta T, Agarwal J, Jain S, Phurailatpam R, Kannan S, Ghosh-Laskar S, Murthy V, Budrukkar A, Dinshaw K, Prabhash K, Chaturvedi P, D'Cruz A. Three-dimensional conformal radiotherapy (3D-CRT) versus intensity modulated radiation therapy (IMRT) in squamous cell carcinoma of the head and neck: a randomized controlled trial. Radiother Oncol. 2012 Sep;104(3):343-8. doi: 10.1016/j.radonc.2012.07.001. Epub 2012 Jul 30. PMID 22853852
- [Background] Xiong H, Liao Z, Liu Z, Xu T, Wang Q, Liu H, Komaki R, Gomez D, Wang LE, Wei Q. ATM polymorphisms predict severe radiation pneumonitis in patients with non-small cell lung cancer treated with definitive radiation therapy. Int J Radiat Oncol Biol Phys. 2013 Mar 15;85(4):1066-73. doi: 10.1016/j.ijrobp.2012.09.024. Epub 2012 Nov 12. PMID 23154078
- [Background] Cheuk IW, Yip SP, Kwong DL, Wu VW. Association of XRCC1 and XRCC3 gene haplotypes with the development of radiation-induced fibrosis in patients with nasopharyngeal carcinoma. Mol Clin Oncol. 2014 Jul;2(4):553-558. doi: 10.3892/mco.2014.276. Epub 2014 Apr 14. PMID 24940494
- [Background] Bray FN, Simmons BJ, Wolfson AH, Nouri K. Acute and Chronic Cutaneous Reactions to Ionizing Radiation Therapy. Dermatol Ther (Heidelb). 2016 Jun;6(2):185-206. doi: 10.1007/s13555-016-0120-y. Epub 2016 Jun 1. PMID 27250839
- [Background] Suarez EM, Knackstedt RJ, Jenrette JM. Significant fibrosis after radiation therapy in a patient with Marfan syndrome. Radiat Oncol J. 2014 Sep;32(3):208-12. doi: 10.3857/roj.2014.32.3.208. Epub 2014 Sep 30. PMID 25324993
- [Background] Nevens D, Duprez F, Daisne JF, Laenen A, De Neve W, Nuyts S. Radiotherapy induced dermatitis is a strong predictor for late fibrosis in head and neck cancer. The development of a predictive model for late fibrosis. Radiother Oncol. 2017 Feb;122(2):212-216. doi: 10.1016/j.radonc.2016.08.013. Epub 2016 Sep 20. PMID 27663951
- [Background] Hamada K, Fujibuchi T, Arakawa H, Yokoyama Y, Yoshida N, Ohura H, Kunitake N, Masuda M, Honda T, Tokuda S, Sasaki M. A novel approach to predict acute radiation dermatitis in patients with head and neck cancer using a model based on Bayesian probability. Phys Med. 2023 Dec;116:103181. doi: 10.1016/j.ejmp.2023.103181. Epub 2023 Nov 24. PMID 38000101
- [Background] Lee TF, Liu YH, Chang CH, Chiu CL, Lin CH, Shao JC, Yen YC, Lin GZ, Yang J, Tseng CD, Fang FM, Chao PJ, Lee SH. Development of a risk prediction model for radiation dermatitis following proton radiotherapy in head and neck cancer using ensemble machine learning. Radiat Oncol. 2024 Jun 24;19(1):78. doi: 10.1186/s13014-024-02470-1. PMID 38915112
- [Background] Bontempo PSM, Meneses AG, Ciol MA, Ferreira EB, Reis PEDD. Instruments and scales for the evaluation of acute radiation dermatitis: A systematic review. Crit Rev Oncol Hematol. 2023 Nov;191:104116. doi: 10.1016/j.critrevonc.2023.104116. Epub 2023 Aug 28. PMID 37648000
- [Background] Noble-Adams R. Radiation-induced skin reactions. 2: Development of a measurement tool. Br J Nurs. 1999 Oct 14-27;8(18):1208-11. doi: 10.12968/bjon.1999.8.18.6490. PMID 10897708
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Background] Huang CJ, Hou MF, Luo KH, Wei SY, Huang MY, Su SJ, Kuo HY, Yuan SS, Chen GS, Hu SC, Chuang HY. RTOG, CTCAE and WHO criteria for acute radiation dermatitis correlate with cutaneous blood flow measurements. Breast. 2015 Jun;24(3):230-6. doi: 10.1016/j.breast.2015.01.008. Epub 2015 Mar 14. PMID 25777626
- [Background] Berthelet E, Truong PT, Musso K, Grant V, Kwan W, Moravan V, Patterson K, Olivotto IA. Preliminary reliability and validity testing of a new Skin Toxicity Assessment Tool (STAT) in breast cancer patients undergoing radiotherapy. Am J Clin Oncol. 2004 Dec;27(6):626-31. doi: 10.1097/01.coc.0000138965.97476.0f. PMID 15577442
- [Background] Aguiar BRL, Ferreira EB, Normando AGC, Mazzeu JF, Assad DX, Guerra ENS, Reis PEDD. Single nucleotide polymorphisms to predict acute radiation dermatitis in breast cancer patients: A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2022 May;173:103651. doi: 10.1016/j.critrevonc.2022.103651. Epub 2022 Mar 15. PMID 35301098
- [Background] Yu J, Huang Y, Liu L, Wang J, Yin J, Huang L, Chen S, Li J, Yuan H, Yang G, Liu W, Wang H, Pei Q, Guo C. Genetic polymorphisms of Wnt/beta-catenin pathway genes are associated with the efficacy and toxicities of radiotherapy in patients with nasopharyngeal carcinoma. Oncotarget. 2016 Dec 13;7(50):82528-82537. doi: 10.18632/oncotarget.12754. PMID 27769064
- [Background] Mumbrekar KD, Bola Sadashiva SR, Kabekkodu SP, Fernandes DJ, Vadhiraja BM, Suga T, Shoji Y, Nakayama F, Imai T, Satyamoorthy K. Genetic Variants in CD44 and MAT1A Confer Susceptibility to Acute Skin Reaction in Breast Cancer Patients Undergoing Radiation Therapy. Int J Radiat Oncol Biol Phys. 2017 Jan 1;97(1):118-127. doi: 10.1016/j.ijrobp.2016.09.017. Epub 2016 Sep 20. PMID 27816361
- [Background] Isomura M, Oya N, Tachiiri S, Kaneyasu Y, Nishimura Y, Akimoto T, Hareyama M, Sugita T, Mitsuhashi N, Yamashita T, Aoki M, Sai H, Hirokawa Y, Sakata K, Karasawa K, Tomida A, Tsuruo T, Miki Y, Noda T, Hiraoka M. IL12RB2 and ABCA1 genes are associated with susceptibility to radiation dermatitis. Clin Cancer Res. 2008 Oct 15;14(20):6683-9. doi: 10.1158/1078-0432.CCR-07-4389. PMID 18927311
- [Background] Aguiar BRL, Ferreira EB, Normando AGC, Dias SDS, Guerra ENS, Reis PED. Potential Single Nucleotide Polymorphisms markers for radiation dermatitis in head and neck cancer patients: a meta-analysis. Strahlenther Onkol. 2024 Jul;200(7):568-582. doi: 10.1007/s00066-024-02237-3. Epub 2024 Apr 26. PMID 38668865
- [Background] De Langhe S, Mulliez T, Veldeman L, Remouchamps V, van Greveling A, Gilsoul M, De Schepper E, De Ruyck K, De Neve W, Thierens H. Factors modifying the risk for developing acute skin toxicity after whole-breast intensity modulated radiotherapy. BMC Cancer. 2014 Sep 25;14:711. doi: 10.1186/1471-2407-14-711. PMID 25252713
- [Background] Ramia P, Bodgi L, Mahmoud D, Mohammad MA, Youssef B, Kopek N, Al-Shamsi H, Dagher M, Abu-Gheida I. Radiation-Induced Fibrosis in Patients with Head and Neck Cancer: A Review of Pathogenesis and Clinical Outcomes. Clin Med Insights Oncol. 2022 Jan 30;16:11795549211036898. doi: 10.1177/11795549211036898. eCollection 2022. PMID 35125900
- [Background] Gosselin T, Ginex PK, Backler C, Bruce SD, Hutton A, Marquez CM, McGee LA, Shaftic AM, Suarez LV, Moriarty KA, Maloney C, Vrabel M, Morgan RL. ONS Guidelines for Cancer Treatment-Related Radiodermatitis. Oncol Nurs Forum. 2020 Nov 1;47(6):654-670. doi: 10.1188/20.ONF.654-670. PMID 33063779
- [Background] Dorr W. Skin and other reactions to radiotherapy--clinical presentation and radiobiology of skin reactions. Front Radiat Ther Oncol. 2006;39:96-101. doi: 10.1159/000090854. No abstract available. PMID 16394673
- [Background] Kyei KA, Daniels J, Pratt-Ainooson F, Anim-Sampong S, Nkansah EO, Amoabeng KA, Antwi WK. Incidence and severity of acute radiation induced toxicities among breast cancer patients treated with adjuvant radiotherapy at a major cancer treatment center in Ghana. Transl Oncol. 2024 Sep;47:102032. doi: 10.1016/j.tranon.2024.102032. Epub 2024 Jun 29. PMID 38945020
- [Background] Eggert MC, Yu NY, Rades D. Radiation Dermatitis and Pneumonitis in Patients Irradiated for Breast Cancer. In Vivo. 2023 Nov-Dec;37(6):2654-2661. doi: 10.21873/invivo.13374. PMID 37905621
- [Background] Bontempo PSM, Ciol MA, Meneses AG, Simino GPR, Ferreira EB, Reis PEDD. Acute radiodermatitis in cancer patients: incidence and severity estimates. Rev Esc Enferm USP. 2021 Apr 16;55:e03676. doi: 10.1590/S1980-220X2019021703676. eCollection 2021. English, Portuguese. PMID 33886907
- [Background] Fijardo M, Kwan JYY, Bissey PA, Citrin DE, Yip KW, Liu FF. The clinical manifestations and molecular pathogenesis of radiation fibrosis. EBioMedicine. 2024 May;103:105089. doi: 10.1016/j.ebiom.2024.105089. Epub 2024 Apr 5. PMID 38579363
- [Background] Xie Y, Hu T, Chen R, Chang H, Wang Q, Cheng J. Predicting acute radiation dermatitis in breast cancer: a prospective cohort study. BMC Cancer. 2023 Jun 12;23(1):537. doi: 10.1186/s12885-023-10821-6. PMID 37308936
- [Background] Kawamura M, Yoshimura M, Asada H, Nakamura M, Matsuo Y, Mizowaki T. A scoring system predicting acute radiation dermatitis in patients with head and neck cancer treated with intensity-modulated radiotherapy. Radiat Oncol. 2019 Jan 21;14(1):14. doi: 10.1186/s13014-019-1215-2. PMID 30665451
- [Background] Tenorio C, de la Mata D, Leyva JAF, Poitevin-Chacon A, Queijeiro MV, Gutierrez GR, Nogueda JC, Cons LCD, Hernandez YB, Sanchez DR, Cruz AAS, Guardado GN, Tomasena MI, Ortiz S, Del Bosque MAS, Garzon LAC, Puch AES, Retif RP, Arceo PRL, Lopez LHB, Baldi CMT. Mexican radiationdermatitis management consensus. Rep Pract Oncol Radiother. 2022 Oct 31;27(5):914-926. doi: 10.5603/RPOR.a2022.0101. eCollection 2022. PMID 36523808
- [Background] Spalek M. Chronic radiation-induced dermatitis: challenges and solutions. Clin Cosmet Investig Dermatol. 2016 Dec 9;9:473-482. doi: 10.2147/CCID.S94320. eCollection 2016. PMID 28003769
- [Background] Wei J, Meng L, Hou X, Qu C, Wang B, Xin Y, Jiang X. Radiation-induced skin reactions: mechanism and treatment. Cancer Manag Res. 2018 Dec 21;11:167-177. doi: 10.2147/CMAR.S188655. eCollection 2019. PMID 30613164
- [Background] Singh M, Alavi A, Wong R, Akita S. Radiodermatitis: A Review of Our Current Understanding. Am J Clin Dermatol. 2016 Jun;17(3):277-92. doi: 10.1007/s40257-016-0186-4. PMID 27021652
- [Background] Behroozian T, Goldshtein D, Ryan Wolf J, van den Hurk C, Finkelstein S, Lam H, Patel P, Kanee L, Lee SF, Chan AW, Wong HCY, Caini S, Mahal S, Kennedy S, Chow E, Bonomo P; Multinational Association of Supportive Care in Cancer (MASCC) Oncodermatology Study Group Radiation Dermatitis Guidelines Working Group. MASCC clinical practice guidelines for the prevention and management of acute radiation dermatitis: part 1) systematic review. EClinicalMedicine. 2023 Mar 27;58:101886. doi: 10.1016/j.eclinm.2023.101886. eCollection 2023 Apr. PMID 37181415